CLINICAL TRIAL: NCT02795195
Title: Phase I/II Trail Evaluating Carbon Ion Radiotherapy (3 GyE Per Fraction) for Salvaging Treatment of Locally Recurrent Nasopharyngeal Carcinoma
Brief Title: Trail Evaluating Carbon Ion Radiotherapy (3 GyE Per Fraction) for Locally Recurrent Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Proton and Heavy Ion Center (Other)
Responsible Party: Principal Investigator, Jiade J. Lu, Professor, Shanghai Proton and Heavy Ion Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPHIC-TR-HNCNS-2015-03
Record Dates: First submitted 2016-06-06; First posted 2016-06-10 (Estimated); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: re-irradiation; carbon ion therapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Heavy Ion Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CIRT Arm (3GyE per fraction) (Experimental): Patients included in this arm were treated with carbon ion radiotherapy with a fraction size of 3GyE.
  Interventions: Radiation: Carbon ion radiotherapy (CIRT)

INTERVENTIONS:
Radiation: Carbon ion radiotherapy (CIRT) — Five dose levels (51GyE, 54GyE, 57GyE, 60GyE, 63GyE) are planned within the Phase I part. And the started dose level will be 54GyE. Daily fraction of 3 GyE will be delivered for all dose levels. After the recommended dose (RD), i.e., maximal tolerated dose, is determined or if the treatments to 63 GyE are safely delivered, the recommended dose (or 63 GyE) will be the prescribed dose in the Phase II part of the study.

SUMMARY:
The purpose of this study is to determine the maximal tolerated dose (MTD) of re-irradiation using carbon ion radiotherapy (CIRT) with the fraction size of 3 gray equivalent (GyE) in the treatment of locally recurrent nasopharyngeal cancer (NPC) and to evaluate the efficacy of such treatment at the MTD. Participants will be treated with CIRT with escalating dose regimens to evaluate the MTD in terms of acute and subacute toxicity observed within 4 months after the completion of CIRT. Once the MTD for locally recurrent NPC is determined, the MTD will be used as the recommended dose to patients fulfilling the inclusion criteria in the Phase II part of the trial.

DETAILED DESCRIPTION:
The purpose of this study is to determine the maximal tolerated dose (MTD) of re-irradiation using carbon ion radiotherapy (CIRT) with the fraction size of 3 GyE in the treatment of locally recurrent nasopharyngeal cancer (NPC) and to evaluate the efficacy of such treatment at the MTD. Participants will be treated with CIRT with escalating dose starting from 54GyE (3GyE/daily fraction) to potentially 63GyE (3GyE/daily fraction) to evaluate the maximal tolerated dose (MTD) in terms of acute and subacute toxicity observed during and within 4 months after the completion of CIRT. The TITE-CRM method is used for the phase I dose escalating part of the trial and approximately 25 patients will be accrued. Once the MTD for locally recurrent NPC is determined, the MTD will be used as the recommended dose to patients fulfilling the inclusion criteria in the Phase II part of the trial. The Phase II part of the trial will be a single stage single arm study.

ELIGIBILITY:
Inclusion Criteria:

* Completed a definitive course of intensity-modulated photon radiation therapy (IMXT) to a total dose of ≥ 66 Gy
* Recurrence diagnosed more than 12 months after the initial course of IMXT
* Age ≥ 18 and < 70 years of age
* Karnofsky Performance Score ≥70
* Willing to accept adequate contraception for women with childbearing potential
* Ability to understand character and individual consequences of the clinical trial
* Willing to sign the written informed consent; Informed consent must be signed before the enrollment in the trial

Exclusion Criteria:

* Presence of distant metastasis
* Technology used other than IMXT (including brachytherapy following IMXT) for the treatment of initial diagnosis of NPC
* Pregnant or lactating women
* Patients who have not yet recovered from acute toxicities of prior therapies
* A diagnosis of malignancy other than carcinoma in situ of the cervix, basal cell carcinoma and squamous cell carcinoma of the skin within the past 5 years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2021-04-22 (Actual); Study Completion 2021-04-22 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 (phase 1) | Within 4 months after the completion of treatment
  The primary objective of phase 1 is to identify the maximum tolerated dose which is defined as the highest dose associated with a probability of dose limiting toxicity <=25%.
Phase 2: Overall survival (OS) | 2 years
  Overall survival (OS) was defined as the time frame from enrollment to the date of death from any cause.

SECONDARY OUTCOMES:
Phase 2: Progression-free survival | 2 years
  Progression-free survival (PFS) was defined as the time frame from enrollment to the date of disease progression or death whichever came first.

CONTACTS AND LOCATIONS:
Overall Officials: Jiade J Lu, MD, Principal Investigator — Shanghai Proton and Heavy Ion Center,Shanghai, SPHIC
Locations (1):
- Shanghai Proton and Heavy Ion Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No